CLINICAL TRIAL: NCT02774902
Title: A Phase 1, Open-Label, Sequential Design Study to Evaluate the Effect of Multiple Oral Doses of Clarithromycin on the Pharmacokinetics of a Single Oral Dose of TAK-438
Brief Title: TAK-438_110 Drug Interaction With Cytochrome P450 3A4 (CYP3A4) Inhibitor Clarithromycin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-438-110; 2010-020813-10 (EudraCT Number); U1111-1181-8324 (Registry Identifier: WHO)
Record Dates: First submitted 2016-05-13; First posted 2016-05-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAK-438 40 mg + Clarithromycin 500 mg (Experimental): TAK-438 40 mg, tablets, orally once on Days 1 and 8 along with clarithromycin 500 mg, tablets, orally twice daily from Days 3 to 9.
  Interventions: Drug: TAK-438; Drug: Clarithromycin

INTERVENTIONS:
Drug: TAK-438 — TAK-438 tablets
Drug: Clarithromycin — Clarithromycin tablets

SUMMARY:
The purpose of this study is to evaluate the effect of multiple oral doses of clarithromycin on the pharmacokinetics of TAK-438 and its metabolites in healthy male adult participants following a single oral dose of TAK-438.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-438. TAK 438 is being tested to assess the effect of multiple oral doses of clarithromycin on the pharmacokinetics of TAK-438.

The study will enroll approximately 16 healthy adult male participants of non-Japanese origin. Participants will be assigned:

* TAK-438 40 mg
* Clarithromycin 500 mg

All participants will be asked to take 2 tablet of TAK-438 20 mg orally, once on Days 1 and 8 along with Clarithromycin 500 mg, tablets, orally twice daily from Days 3 to 9.

This single center trial will be conducted in Europe. The overall time to participate in this study is maximum of 44 days. Participants will be confined to site for 10 days, and a final visit after 4 days after discharge from the unit for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Is a healthy adult male participant, of non-Japanese origin.
4. Is aged 18 to 45 years, inclusive, at the time of informed consent and first study medication dose.
5. Weighs at least 45 kg and has a body mass index (BMI) between 18 and 30 kg/m^2, inclusive at Screening.
6. A male participant who is sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after last dose.
7. Has clinical laboratory evaluations (including clinical chemistry, hematology, and urinalysis), within the reference range for the testing laboratory. Participants with evaluations outside the reference range that are deemed not clinically significant by the investigator may be included at investigator discretion unless these are specifically identified in the exclusion criteria.
8. Is willing to abstain from caffeine and alcohol from 72 hours before first dose (Day 1) until the Follow-up call.
9. Is willing to abstain from strenuous exercise from 72 hours before first dose (Day 1) until the Follow-up call.
10. Is willing to provide a sample for pharmacogenomic analysis.

Exclusion Criteria:

1. Has received any investigational compound within 90 days prior to the first dose on Day 1.
2. Has received TAK-438 in a previous clinical study or as a therapeutic agent.
3. Is an immediate family member, study site employee, or in a dependant relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
4. Has a known hypersensitivity or allergies to clarithromycin or any associated excipients.
5. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 5 years prior to the Screening Visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
6. Has taken or is required to take any excluded medication.
7. Intends to donate sperm during the course of this study or for 12 weeks thereafter.
8. Has evidence of current cardiovascular, central nervous system, hepatic, hematopoietic disease, renal dysfunction, metabolic or endocrine dysfunction, serious allergy, asthma hypoxemia, hypertension, seizures, or allergic skin rash. There is any finding in the participant's medical history, physical examination, or safety laboratory tests giving reasonable suspicion of a disease that would contraindicate taking TAK-438, or a similar drug in the same class, or clarithromycin, or that might interfere with the conduct of the study. This includes, but is not limited to, peptic ulcer disease, seizure disorders, and cardiac arrhythmias.
9. Has a history or clinical manifestations of significant symptomatic, gastroesophageal reflux disease (GERD), erosive esophagitis (EE), duodenal ulcer, gastric ulcer, dyspepsia, Barrett esophagus (BE), or Zollinger-Ellison syndrome.
10. Has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (ie, a history of malabsorption, esophageal reflux, peptic ulcer disease, EE frequent [more than once per week], occurrence of heartburn, or any surgical intervention [eg, cholecystectomy]).
11. Has a history of cancer, except basal cell carcinoma that has been in remission for at least 5 years prior to Day 1.
12. Has a positive test result for hepatitis A, hepatitis B surface antigen, antibody to hepatitis C virus, or human immunodeficiency virus at Screening.
13. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 6 weeks prior to Check-in Day -1. Urine test is positive at Screening or Check-in (Day -1).
14. Has a positive alcohol breath test at the Screening or Check-in (Day -1).
15. Has confirmed positive result for drugs of abuse at the Screening Visit or Check-in (Day -1).
16. Has abnormal Screening or Day -1 laboratory values that suggest a clinically significant underlying disease or participant with the following laboratory abnormalities: has an alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level which exceeds 3*upper limit of normal (ULN) set by the testing laboratory at the Screening Visit or Check-in (Day -1).
17. Has poor peripheral venous access.
18. Has donated or lost 450 mL or more of his or her blood volume (including plasmapheresis), or had a transfusion of any blood product within 90 days prior to Day 1.
19. Is unable to understand verbal or written English or any other language for which a certified translation of the informed consent and other material supplied for completion by participant is available.
20. Has a Screening or Check-in (Day -1) abnormal (clinically significant) electrocardiogram (ECG). Entry of any participant with an abnormal (not clinically significant) ECG must be approved, and documented by signature by the principal investigator.
21. Has a marked baseline prolongation of QT/QTc interval (eg, repeated demonstration of a QTc interval >450 ms) on ECG at the Screening Visit.
22. Has a history of clinically significant inflammatory disease or allergy (eg, hay fever [hay fever sufferers who do not require medication may be permitted], asthma, eczema), autoimmune disease (eg, psoriasis, lupus), or history of chronic respiratory disease (eg, emphysema or chronic obstructive pulmonary disease).
23. Has a history of additional risk factors for torsades de pointes (eg, heart failure, hypokalemia, family history of Long QT Syndrome).
24. Is considered by the investigator, for any reason, to be an unsuitable candidate for participating in this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration for TAK-438 and TAK-438 Metabolites (M-I, M-II, M-III, M-IV-Sul) | Days 1 and 8 pre-dose and at multiple timepoints (up to 48 hours) post-dose
AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-438 and TAK-438 Metabolites (M-I, M-II, M-III, M-IV-Sul) | Days 1 and 8 pre-dose and at multiple timepoints (up to 48 hours) post-dose
AUC∞: Area Under the Plasma Concentration-time Curve from Time 0 to Infinity for TAK-438 and TAK-438 Metabolites (M-I, M-II, M-III, M-IV-Sul) | Days 1 and 8 pre-dose and at multiple timepoints (up to 48 hours) post-dose
AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours Postdose for TAK-438 and TAK-438 Metabolites (M-I, M-II, M-III, M-IV-Sul) | Days 1 and 8 pre-dose and at multiple timepoints (up to 48 hours) post-dose

SECONDARY OUTCOMES:
Ratio of TAK-438 Metabolites Cmax to TAK-438 Cmax | Days 1 and 8 pre-dose and at multiple timepoints (up to 48 hours) post-dose
Ratio of TAK-438 Metabolites AUClast to TAK-438 AUClast | Days 1 and 8 pre-dose and at multiple timepoints (up to 48 hours) post-dose
Ratio of TAK-438 Metabolites AUC∞ to TAK-438 AUC∞ | Days 1 and 8 pre-dose and at multiple timepoints (up to 48 hours) post-dose
Ratio of TAK-438 Metabolites AUC(0-24) to TAK-438 AUC(0-24) | Days 1 and 8 pre-dose and at multiple timepoints (up to 48 hours) post-dose
Predose Observed Plasma Concentration of Clarithromycin | Days 3 to 9 pre-dose (-1 hours [1 hour before TAK-438 dosing]) and (11 hours [11 hours after TAK 438 dosing])
Percentage of Participants who Experience at Least One Treatment Emergent Adverse Event (TEAE) | Day 1 until Day 14 or early termination
Percentage of Participants With Markedly Abnormal Laboratory Values | Screening (Days -28 to -2) up to Day 10
Percentage of Participants With Markedly Abnormal Vital Sign Measurements at Least Once Post-dose | Screening (Days -28 to -2) up to Day 10
Percentage of Participants With Markedly Abnormal Safety Electrocardiogram (ECG) Parameters at Least Once Post-dose | Screening (Days -28 to -2) up to Day 10
Percentage of Participants With Clinical Significant Change in Physical Examination | Screening (Days -28 to -2) up to Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda

REFERENCES:
- [Derived] Jenkins H, Jenkins R, Patat A. Effect of Multiple Oral Doses of the Potent CYP3A4 Inhibitor Clarithromycin on the Pharmacokinetics of a Single Oral Dose of Vonoprazan: A Phase I, Open-Label, Sequential Design Study. Clin Drug Investig. 2017 Mar;37(3):311-316. doi: 10.1007/s40261-016-0488-6. PMID 27928738